CLINICAL TRIAL: NCT03150524
Title: RCVS: The Rational Approach to Diagnosis and Treatment
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Failure to recruit patients meeting inclusion criteria.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00130191
Record Dates: First submitted 2017-05-08; First posted 2017-05-12 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Reversible Cerebral Vasoconstriction Syndrome
Keywords: stroke; RCVS
MeSH Terms: conditions — Stroke | interventions — Nimodipine; Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nimodipine (Active Comparator): Patients in group one will receive short-acting nimodipine every 4 hours.
  Interventions: Diagnostic Test: TCD- cerebral blood flow velocities; Behavioral: Headache pain score; Other: Neurological examination; Diagnostic Test: Repeat Neuroimaging; Drug: Nimodipine
- Verapamil ER (Active Comparator): Patients in group two will receive long-acting verapamil every 12 hours.
  Interventions: Diagnostic Test: TCD- cerebral blood flow velocities; Behavioral: Headache pain score; Other: Neurological examination; Diagnostic Test: Repeat Neuroimaging; Drug: Verapamil ER

INTERVENTIONS:
Diagnostic Test: TCD- cerebral blood flow velocities — Participants will undergo daily TCD for monitoring of cerebral blood flow.
Behavioral: Headache pain score — Participants will be evaluated by nurses for headache frequency and severity every shift.
Other: Neurological examination — Patients will be examined routinely for evidence of neurological improvement/decline and/or evidence of a complication such as stroke or hemorrhage.
Diagnostic Test: Repeat Neuroimaging — All patients will also be seen at 90 days (+/- 30 days) and administered a headache diary, repeat neuroimaging, and neurological examination.
Drug: Nimodipine — Participants will be administered nimodipine every 4 hours.
  Arms: Nimodipine
Drug: Verapamil ER — Participants will be administered long acting verapamil every 12 hours.
  Arms: Verapamil ER

SUMMARY:
This is a randomized clinical trial of short-acting nimodipine versus twice daily extended release verapamil to treat patients presenting with Reversible Cerebral Vasoconstriction Syndrome (RCVS).

DETAILED DESCRIPTION:
Patients greater than 18 years of age presenting with clinical signs and symptoms consistent with RCVS (see inclusion criteria) will be enrolled. Neuroimaging (CT, Magnetic Resonance (MR), or 4 vessel angiogram) will be obtained along with a baseline transcranial doppler ultrasound (TCD). They will subsequently be randomized to receive nimodipine (every 4 hours) or extended release verapamil (twice daily). Mean cerebral blood flow velocities will be followed for reduction or normalization on daily TCD and medication dosing adjusted appropriately. Patients will be followed 90 days post-discharge at which time they will undergo repeat neuroimaging to confirm resolution of vascular abnormalities and repeat evaluation. To determine effectiveness, the investigators will evaluate both short-term (surrogate) in-hospital outcomes and long-term outcomes. Reduction of TCD velocities and headache severity will serve as our short-term surrogate outcomes; however, need for additional medications, blood pressure, new/recurrent stroke/Intracranial Hemorrhage (ICH) will also be evaluated along with modified Rankin score (mRS) on discharge, length of stay, and discharge disposition. At 90 days, the investigators will also assess headache control along with mRS.. Adverse events and their relation to the treatment arms will be assessed, and adherence to the medications will be evaluated.

ELIGIBILITY:
Patients 18 years of age or greater meeting the following inclusion criteria adapted from Singhal and colleagues 2 will be included:

1. presentation consistent with RCVS :

* acute thunderclap/severe headache and

  **supporting clinical features should prompt increased clinical suspicion (eg., potential medication trigger, recent pregnancy, migraine history)**
* evidence of beading/elevated velocities on imaging (Transcranial Doppler (TCD), angiogram, Computer Tomography Angiogram (CTA), MRA) and
* reversibility (by 90 days)-will not be required for inclusion but will be retrospectively adjudicated

Participants will be excluded from the study if they are:

* unable to consent AND no family present to consent, or
* have presence of aneurysmal, traumatic, or mesencephalic Subarachnoid Hemorrhage (SAH), or
* have presence of other supported diagnosis (eg., vasculitis- inflammatory lumbar puncture) or
* are currently pregnant or
* the use of nimodipine or verapamil is contraindicated for any reason (eg., allergy, breast feeding) or
* have limited TCD sonographic window

  * stroke or ICH/SAH on presentation will not be a contraindication to inclusion in the trial **

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Peak TCD velocities | daily from admission to discharge (approx 5-7 days)
  Peak mean Cerebral Blood Flow velocity (CBFV) in anterior circulation vessels (MCA/Anterior Cerebral Artery (ACA)/Posterior Cerebral Artery (PCA)/internal carotid)
Duration of elevated TCD velocities | daily from admission to discharge (approx 5-7 days)
  Duration of elevated velocity (number of days from presentation to normalization/reduction)
Normalization of TCD velocities | daily from admission to discharge (approx 5-7 days)
  Normalization/reduction of velocity (yes/no)

SECONDARY OUTCOMES:
Peak pain score | every 8 hours while hospitalized (approx 5-7 days) and at 90 day follow-up
  Peak pain score- Likert scale evaluating headache: 0-10 points
Days to pain resolution | every 8 hours while hospitalized (approx 5-7 days) and at 90 day follow-up
  Number of days to resolution
New or recurrent stroke/hemorrhage | daily through hospitalization (approx 5-7 days)
  evaluated by neurological examinations and confirmed by imaging
Modified Rankin Scale | on hospital discharge and at 90 day follow-up
  functional outcome scale based on mobility and ability to perform activities of daily living- scale 0-6 points (0-2 considered good outcome)
Repeat neuroimaging | at 90 day follow-up
  repeat neuroimaging to confirm reversibility of vasculopathy
Medication compliance | daily throughout hospitalization (approx 5-7 days) and at 90 day follow-up
  ability to tolerate and adhere to medication

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth B Marsh, MD, Principal Investigator — Johns Hopkins University; Rafael H Llinas, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singhal AB, Hajj-Ali RA, Topcuoglu MA, Fok J, Bena J, Yang D, Calabrese LH. Reversible cerebral vasoconstriction syndromes: analysis of 139 cases. Arch Neurol. 2011 Aug;68(8):1005-12. doi: 10.1001/archneurol.2011.68. Epub 2011 Apr 11. PMID 21482916
- [Background] Marsh EB, Ziai WC, Llinas RH. The Need for a Rational Approach to Vasoconstrictive Syndromes: Transcranial Doppler and Calcium Channel Blockade in Reversible Cerebral Vasoconstriction Syndrome. Case Rep Neurol. 2016 Jul 29;8(2):161-171. doi: 10.1159/000447626. eCollection 2016 May-Aug. PMID 27721780
- See also: Johns Hopkins School of Medicine Stroke Division Website — http://www.hopkinsmedicine.org/neurology_neurosurgery/centers_clinics/cerebrovascular/stroke/team.html